CLINICAL TRIAL: NCT03069508
Title: A Phase IIa, Open Label Pilot Study of Clemizole Hydrochloride Given Orally Thrice a Day, for Subjects With Hepatocellular Carcinoma That Are Either Awaiting Transplantation or Have an Unresectable Lesion
Brief Title: Clemizole HCl for Subjects With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eiger Group International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIG-234
Record Dates: First submitted 2017-02-14; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — clemizole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 200 mg TID (Experimental): 200 mg clemizole hydrochloride will be administered orally thrice a day for 24 weeks.
  Interventions: Drug: Clemizole Hydrochloride
- 300 mg TID (Experimental): 300 mg clemizole hydrochloride will be administered orally thrice a day for 24 weeks.
  Interventions: Drug: Clemizole Hydrochloride
- 400 mg TID (Experimental): 400 mg clemizole hydrochloride will be administered orally thrice a day for 24 weeks.
  Interventions: Drug: Clemizole Hydrochloride
- 500 mg TID (Experimental): 500 mg clemizole hydrochloride will be administered orally thrice a day for 24 weeks.
  Interventions: Drug: Clemizole Hydrochloride

INTERVENTIONS:
Drug: Clemizole Hydrochloride — Clemizole Hydrochloride will be administered orally for up to 24 weeks
  Other Names: Clemizole

SUMMARY:
This study is a phase IIa open label pilot study of up to six months treatment with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 vs. 500 mg mg) given orally TID to subjects with hepatocellular carcinoma that are either awaiting transplantation or have an unresectable lesion.

DETAILED DESCRIPTION:
The primary objectives of the study are to:

* Evaluate the safety and tolerability of up to six months of treatment with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg TID by mouth) in subjects diagnosed with hepatocellular carcinoma that are either awaiting transplantation or have an unresectable lesion.
* Evaluate the overall tumor response according to radiologic assessments of stable disease, complete response (CR), partial response (PR), or minor response (MR), as defined by Response Evaluation Criteria in Solid Tumors (RECIST), associated with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)
* Evaluate the pharmacokinetic (PK) activity of clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)

The secondary objectives of the study are to:

• Evaluate the duration of response, time to progression, duration of stable disease (SD), and overall survival associated with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, at least 18 years of age.
2. Subjects should have a diagnosis (histologically proven) of hepatocellular carcinoma (that is measurable on CT or MR with contrast) and are either awaiting transplantation or have an unresectable lesion for which they have not received prior experimental systemic treatments for HCC and no additional therapy is planned.
3. Eastern Cooperative Oncology Group performance status of 2 or less.
4. Child-Pugh (CP) score of A or B.
5. Life expectancy of at least 12 weeks.
6. Elevated alphafetoprotein (AFP) level .
7. Adequate hematologic (platelet count, ≥60 ; hemoglobin, ≥8.5 g per deciliter; and prothrombin time international normalized ratio, ≤2.3; or prothrombin time, ≤6 seconds above control), hepatic (albumin, ≥2.8 g per deciliter; total bilirubin, ≤3 mg per deciliter [51.3 μmol per liter]; and alanine aminotransferase and aspartate aminotransferase, ≤5 times the upper limit of the normal range), and renal (serum creatinine, ≤1.5 times the upper limit of the normal range) function.
8. Electrocardiogram (ECG) showing no acute ischemia or clinically significant abnormality and a QT/QTc interval <450 milliseconds for males or <470 milliseconds for females using Bazett's correction (QTc =QT/RR0.5;ICH Guidance E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs)
9. Females of childbearing potential (intact uterus and within one year since the last menstrual period) should be non-lactating and have a negative serum pregnancy test. In addition, all subjects (male and female) and their sexually active partners should agree to use one of the following acceptable birth control methods throughout the study:

   1. surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) six month minimum
   2. IUD in place for at least three months
   3. barrier methods (condom or diaphragm) with spermicide
   4. surgical sterilization of the partner (vasectomy for six months)
   5. hormonal contraceptives for at least three months prior to the first dose of study drug
10. Willing and able to comply with study procedures and provide written informed consent

Exclusion Criteria:

1. Participation in a clinical trial with or use of any investigational agent within 30 days of Study Visit 1
2. Patients co-infected with HIV
3. Patients with screening tests positive for anti-HIV Ab
4. Patients with tumors of mixed histology or fibrolamellar variant,
5. Pregnant or lactating women,
6. Patients requiring systemic anticancer therapy, or biologic-response modifiers
7. Medical/psychological/social problems that might affect study participation or evaluations
8. Eating disorder or alcohol abuse within the past two years, excessive alcohol intake (>20 g per day for females (1.5 standard alcohol drinks) or >30 g per day for males (2.0 standard alcohol drinks) (a standard drink contains 14 g of alcohol: 12 oz of beer, 5 oz of wine or 1.5 oz of spirits) (1.0 fluid oz (US) = 29.57 mL) or if in the opinion of the investigator, an alcohol use pattern that will interfere with study conduct
9. Drug abuse within the last six months
10. Patients with absolute neutrophil count (ANC) <1500 cells/mm3;
11. Abnormal TSH, T4 or T3
12. History or clinical evidence of any of the following:

    1. variceal bleeding, difficult to treat ascites, hepatic encephalopathy, CTP score >8,
    2. immunologically mediated disease (e.g, rheumatoid arthritis, inflammatory bowel disease, severe psoriasis, systemic lupus erythematosus) requiring more than intermittent non-steroidal anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids (inhaled asthma medications are allowed)
    3. significant or unstable cardiac disease (e.g., angina, congestive heart failure, uncontrolled hypertension, history of arrhythmia)
    4. chronic pulmonary disease (e.g., chronic obstructive pulmonary disease) associated with functional impairment
    5. severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization
13. Patients with a body mass index of >30 kg/m2
14. Chronic use of concomitant drugs known to prolong the QT interval (See Appendix E)
15. Concomitant use of immunosuppressive or immune modulating agents
16. Patients with any serious condition that, in the opinion of the investigator, would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed or increase the risk to the subject of participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Number of recorded adverse events at six months
  Safety and tolerability of up to six months of treatment with clemizole hydrochloride thrice daily by mouth in subjects diagnosed with hepatocellular carcinoma that are either awaiting transplantation or have an unresectable lesion, determined by the number of participants with abnormal laboratory values and/or adverse events that are related to treatment
Overall tumor response according to radiologic assessments associated with clemizole HCl. | Change from baseline up to 24 weeks
  Number of participants with stable disease, complete response (CR), partial response (PR), or minor response (MR), as defined by Response Evaluation Criteria in Solid Tumors (RECIST), associated with clemizole HCl.
AUC Pharmacokinetic (PK) assessment of clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg by mouth) | 0-pre-dose, post dose: 15 min, 30 min, 60 min, 90 min, 2 hours, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours post oral administration of clemizole HCl for those subjects participating in the PK portion of this trial
  Area under the plasma concentration versus time curve (AUC) of clemizole HCl following oral administration of 200 mg vs. 300 mg vs. 400 mg vs. 500 mg.
Cmax Pharmacokinetic (PK) assessment of clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg by mouth) | 0-pre-dose, post dose: 15 min, 30 min, 60 min, 90 min, 2 hours, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours post oral administration of clemizole HCl for those subjects participating in the PK portion of this trial
  Peak plasma concentration (Cmax) of clemizole HCl following oral administration of 200 mg vs. 300 mg vs. 400 mg vs. 500 mg.

SECONDARY OUTCOMES:
Duration of response associated with clemizole hydrochloride | First administration of study drug until progressive disease in patients with objective responses up to 24 weeks.
  Duration of response associated with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)
Time to progression associated with clemizole hydrochloride | First administration of study drug until progressive disease up to 24 weeks.
  Time to progression associated with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)
Duration of stable disease associated with clemizole hydrochloride | First day of receiving clemizole until progressive disease or response up to 24 weeks.
  Duration of stable disease associated with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)
Overall survival associated with clemizole hydrochloride | First day of receiving study medication to death up to 24 weeks.
  Overall survival associated with clemizole hydrochloride (200 mg vs. 300 mg vs. 400 mg vs. 500 mg, TID by mouth)

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Yurdaydin, MD, Principal Investigator — University of Ankara
Locations (1):
- University of Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No